CLINICAL TRIAL: NCT06157749
Title: Validity and Reliability of a Smartphone Application for Gait Assessment
Brief Title: Gait Assessment Via Telephone Application
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 93402A830
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Health, Subjective
Keywords: 3D Computerized Gait Analysis; Gait-Analyzer; Gait Analysis; Smartphone Application
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D Computerized Gait Analysis: The gait analysis will be conducted through 3D computerized gait analysis.
  Interventions: Other: Gait analysis
- Gait-Analyzer: The gait analysis will be performed using a smartphone application called Gait-Analyzer.
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — It will be carried out on a 10-meter flat surface, with the participant walking at normal walking speed.

SUMMARY:
The evaluation of human gait is a crucial component of the clinical assessment and decision-making process. The gold standard in gait analysis is computerized gait analysis, which allows for three-dimensional digital data acquisition through computers (3D Computerized Gait Analysis). However, this technology is not readily accessible in routine analyses, as it proves to be a time-consuming and expensive endeavor in terms of infrastructure and human resources. The utilization of smartphones in clinical applications is on the rise, facilitated by the increasing accessibility of low-cost or free "applications," thereby addressing the limitations associated with traditional gait analysis methods. The Gait-Analyzer application is among the mentioned applications. However, in the literature, no evidence has been found regarding the validity and reliability of Gait-Analyzer application compared to the gold standard 3D computerized gait analysis systems within the context of gait analyses.

The aim of this study is to comparatively examine the effectiveness of the Gait-Analyzer smartphone application with established 3D Computerized Gait Analysis systems, which have proven validity and reliability in gait analyses. Through this research, the study intends to elucidate the validity and reliability of spatiotemporal parameters of walking within the Gait-Analyzer smartphone application.

DETAILED DESCRIPTION:
Voluntary healthy participants will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. 3D Computerized Gait Analysis will be applied to one group first, and Gait-Analyzer smarthphone application will be applied to the other group first.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 26 years.
* Body Mass Index (BMI) within normal limits (18.5-24.9 kg/m2)

Exclusion Criteria:

* Presence of lower extremity rotational problems (such as high femoral anteversion, internal tibial torsion, metatarsus adductus).
* History of Botulinum Toxin Type A (BoNT-A) application or surgery within the last 6 months.
* History of lower extremity injury within the last 6 months.
* Leg length discrepancy.
* Presence of third-degree pes planus.
* Any neurological, rheumatic, musculoskeletal, metabolic, or connective tissue diseases.
* History of pain, deformity, or surgery related to the vertebral column and upper extremities.
* Presence of cognitive, mental, and/or severe psychiatric disorders

Ages: 18 Years to 26 Years | Sex: All
Age Groups: Adult
Study Population: Volunteers willing to participate in the study and who meet the inclusion criteria of being healthy
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Three-Dimensional Computerized Gait Analysis | change from baseline at first week
  Reflective markers are placed on specific anatomical points to record varying joint angles throughout the walking cycle. Patients walk a distance of 9-10 meters, capturing records of their walking patterns and speed in everyday life, either barefoot or using assistive walking devices.
Gait-Analyzer | change from baseline at first week
  Gait-Analyzer is a mobile application for smartphones capable of real-time analysis of walking parameters. Using a smartphone with an Android processor and the "Gait Analyzer" application, directly attached to the participants' lumbar spine (nearest to L5) with a waist belt, participants will be instructed to complete 6 laps (12 forward and backward walks) on a 10-meter walking path.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Erekdağ, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Acibadem Mehmet Ali Aydinlar University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Stuberg WA, Colerick VL, Blanke DJ, Bruce W. Comparison of a clinical gait analysis method using videography and temporal-distance measures with 16-mm cinematography. Phys Ther. 1988 Aug;68(8):1221-5. PMID 3399519
- [Background] Norris BS, Olson SL. Concurrent validity and reliability of two-dimensional video analysis of hip and knee joint motion during mechanical lifting. Physiother Theory Pract. 2011 Oct;27(7):521-30. doi: 10.3109/09593985.2010.533745. Epub 2011 May 15. PMID 21568816
- [Background] Finkbiner MJ, Gaina KM, McRandall MC, Wolf MM, Pardo VM, Reid K, Adams B, Galen SS. Video Movement Analysis Using Smartphones (ViMAS): A Pilot Study. J Vis Exp. 2017 Mar 14;(121):54659. doi: 10.3791/54659. PMID 28362382
- [Background] Kelly M, Jones P, Wuebbles R, Lugade V, Cipriani D, Murray NG. A novel smartphone application is reliable for repeat administration and comparable to the Tekscan Strideway for spatiotemporal gait. Measurement (Lond). 2022 Mar 31;192:110882. doi: 10.1016/j.measurement.2022.110882. Epub 2022 Feb 11. PMID 35369360